CLINICAL TRIAL: NCT02734225
Title: Valoración de la Puesta en Marcha en Artroplastias Totales de Rodilla Mediante un Trabajo Postural en Plataforma Dinamometrica
Brief Title: Influences of Balance Training With a Dynamometric Platform in Total Knee Arthroplasty
Acronym: TKA_DP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Instituto de Investigacion Sanitaria INCLIVA (Other)
Responsible Party: Principal Investigator, Sergio Roig Casasus, Dr., University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DP_Balance_TKA
Record Dates: First submitted 2016-03-02; First posted 2016-04-12 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Knee Osteoarthritis
Keywords: total knee replacement; total knee arthroplasty; rehabilitation; physical therapy; balance
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Recovery of Function

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- EXPERIMENTAL (Experimental): Functional recovery Balance training
  Interventions: Other: Functional Recovery; Other: Balance Training; Other: Dynamometric Platform Training
- CONTROL (Active Comparator): Functional recovery Balance training Dynamometric Platform training
  Interventions: Other: Functional Recovery; Other: Balance Training

INTERVENTIONS:
Other: Functional Recovery — Rehabilitation protocol based on muscle strengthening with isometric, isotonic and counter-resistance with progressive load exercises. Intervention consisted of warm-up phase with passive, active-assisted and active movements, and a work-out phase
Other: Balance Training — Balance and proprioception training using parallel bars, unstable plates, ramps and stairs
Other: Dynamometric Platform Training — Stability tests, weight changes and stability limits, performing both anterior-posterior and medial-lateral movements simultaneously in some cases
  Arms: EXPERIMENTAL

SUMMARY:
Knee osteoarthritis produces degeneration and joint wear that greatly affects the patient's proprioceptive system increasing instability. After total knee arthroplasty intervention, it is recommended that the patient performs a rehabilitation procedure to minimize deficits caused by surgery. In this job it is essential to insist on the importance of recovering balance after total knee arthroplasty intervention, and assess a specifically designed protocol to restore its function. An intervention which includes a dynamometric platform as a training method was proposed. The randomized clinical trial compared a control group that performed balance exercises on parallel bars, unstable plates, ramps and stairs against an experimental group that included dynamometric platforms training as a differentiator.

ELIGIBILITY:
Inclusion Criteria:

* Age between 65 and 85.
* Subjects with knee osteoarthritis that have not been operated before.
* Patients operated with the same total replacement prosthesis.
* Patients operated with the same surgical procedure.
* Time before intervention over 4 weeks.
* Time to start rehabilitation after surgery must be less than 4 weeks.
* The Result in Berg scale must be greater than 21, indicating a medium-low risk of falling.
* the Result of the Mini-Mental State Examination must be equal or greater than 20, which means they do not have moderate or severe cognitive impairment.
* Once the informed consent is read and explained, patients must accept and agree to participate in the study.

Exclusion Criteria:

* Patient does no accept sign the informed consent.
* Patient with morphological alterations hip or ankle (also knee).
* Patient that presents knee flexion out of the range between 70 ° and -20 ° because of the risk posed to suffer a fall.
* Patient with suspected deep vein thrombosis.
* Patient with post-surgical infection of the operated knee.
* Patient with psychiatric disorders: depression, anxious syndrome, etc.
* Patient with pathology of central origin (i.e. cerebellar) that could interfere with the results of the test of balance or strength
* Patient with vestibular pathology that could interfere with the results of the test of balance

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 69 (Actual)
Dates: Start 2009-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | Change from baseline (two weeks after intervention) to after four weeks of training
  Balance among older people with impairment in balance function by assessing the performance of functional tasks from the total score achieved in the 14 items test

SECONDARY OUTCOMES:
Functional Reach (cm) | Change from baseline (two weeks after intervention) to after four weeks of training
  Assesses a patient's stability by measuring the maximum distance an individual can reach forward while standing in a fixed position
Timed Up and Go Test (s) | Change from baseline (two weeks after intervention) to after four weeks of training
  Dynamic balance assessment. Also points at the risk of falling. Time of getting up from a chair, walk three meters, come back and sit again, measured in seconds
Romberg Tests | Change from baseline (two weeks after intervention) to after four weeks of training
  Total score achieved with open and closed eyes and on firm surface
Knee Range of Mobility (º) | Change from baseline (two weeks after intervention) to after four weeks of training
  Knee Range of Mobility (Flexion, Extension) in degrees
Kendall and Lovet scale | Change from baseline (two weeks after intervention) to after four weeks of training
  Muscle Balance estimated with with Kendall and Lovet scale (score from 0 to 5)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Roig-Casasús, Dr, Principal Investigator — University of Valencia

IPD SHARING:
Plan to Share IPD: Undecided